CLINICAL TRIAL: NCT01718873
Title: Randomized Phase 3 Study on the Optimization of Bevacizumab With mFOLFOX/mOXXEL in the Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Optimization of Bevacizumab Scheduling With Chemotherapy for Metastatic Colorectal Cancer
Acronym: OBELICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBELICS; 2011-004997-27 (EudraCT Number)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2021-10

CONDITIONS: Colorectal Cancer
Keywords: metastatic; stage IV
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab before chemotherapy (Experimental): Bevacizumab administered 4 days before each cycle of chemotherapy containing oxaliplatin (mFOLFOX-6 / mOXXEL)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: levo-folinic acid; Drug: 5-fluorouracil; Drug: Capecitabine
- bevacizumab with chemotherapy (Active Comparator): Bevacizumab administered on the first day of each cycle of chemotherapy containing oxaliplatin (mFOLFOX-6 / mOXXEL)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: levo-folinic acid; Drug: 5-fluorouracil; Drug: Capecitabine

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg every 2 weeks for up to 24 weeks. After 24 weeks, those patients without disease progression will receive bevacizumab 7.5 mg/kg every 3 weeks until progression of disease or unacceptable toxicity.
  Other Names: Avastin
Drug: Oxaliplatin — 85mg/m2 IV every 2 weeks for up to 24 weeks
  Other Names: Eloxatin
Drug: levo-folinic acid — 200 mg/m2 IV before 5-fluorouracil infusion, every 2 weeks up to 24 weeks
  Other Names: Lederfolin
Drug: 5-fluorouracil — 400 mg/m2 IV bolus followed by 2400 mg/m2 IV infusion over 46 hours, every 2 weeks for up to 24 weeks (given in mFOLFOX-6 schedule)
  Other Names: Fluorouracil
Drug: Capecitabine — 1000mg/m2 by mouth, twice a day for 10 days, every 2 weeks for up to 24 weeks(given in mOXXEL schedule)
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to evaluate if giving bevacizumab prior to chemotherapy compared to giving bevacizumab at the same time as chemotherapy improves patient overall response to treatment.

DETAILED DESCRIPTION:
OBELICS is a two-arm phase 3 trial comparing in mCRC patients (1:1): concurrent administration of bevacizumab in combination with modified FOLFOX-6 regimen (mFOLFOX-6) or modified OXXEL regimen (mOXXEL), in which bevacizumab is administered the same day as oxaliplatin, (standard arm); and sequential administration of bevacizumab with the same chemotherapeutic regimens, in which bevacizumab is administered 4 days before oxaliplatin at each cycle (experimental arm) Oxaliplatin regimen (mFOLFOX/mOXXEL) is chosen according to local clinical practice at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of colorectal adenoma carcinoma
* Stage IV disease
* Presence of at least one measurable target lesion (according to RECIST), and not previously radiated.
* Age ≥ 18 e ≤ 75 years
* ECOG Performance status 0-1
* Life expectancy >3 months
* Adequate recovery from surgery, with at least 28 days from surgery to date of pre-study biopsy.
* Adequate contraception for male and female patients of child bearing potential
* informed consent

Exclusion Criteria:

* More than one previous line of therapy for metastatic disease
* Prior treatment with bevacizumab or oxaliplatin (previous treatment with irinotecan,, cetuximab, fluoropyrimidine, folic acid are permitted)
* Primary tumor that is stenosing and/or that infiltrates the entire thickness of the intestinal wall
* Regular use of NSAIDs or aspirin
* Bleeding disorders or coagulopathy
* Concurrent anticoagulant therapy
* Suspected or cerebral metastases (to verify in the presence of symptoms)
* Neutrophils < 2000 / mm3, platelets < 100,000 / mm3, hemoglobin < 9g/dl
* Creatinine > 1.5 times the upper normal limit
* GOT and/or GPT > 2.5 times the upper normal limit, bilirubin > 1.5 times the upper normal limit in absence of liver metastases
* GOT and/or GPT > 5 times the upper normal limit, bilirubin > 3 times the upper normal limit in presence of liver metastases
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal and squamous cell carcinoma or cervical cancer in situ
* Congestive heart failure, ischemic coronary events within past 12 months, uncontrolled cardiac arrhythmia
* Uncontrolled hypertension
* Active or uncontrolled infection
* Any concomitant condition that, in the investigator's opinion, would contraindicate the use of any of the study drugs
* Pregnancy or lactation
* Central nervous system disorders or peripheral neuropathy > grade 1 (CTCAE v. 4.0)
* Inability to comply with follow up procedures of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Italy

REFERENCES:
- [Derived] Avallone A, Piccirillo MC, Nasti G, Rosati G, Carlomagno C, Di Gennaro E, Romano C, Tatangelo F, Granata V, Cassata A, Silvestro L, De Stefano A, Aloj L, Vicario V, Nappi A, Leone A, Bilancia D, Arenare L, Petrillo A, Lastoria S, Gallo C, Botti G, Delrio P, Izzo F, Perrone F, Budillon A. Effect of Bevacizumab in Combination With Standard Oxaliplatin-Based Regimens in Patients With Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2118475. doi: 10.1001/jamanetworkopen.2021.18475. PMID 34309665
- [Derived] Avallone A, Piccirillo MC, Aloj L, Nasti G, Delrio P, Izzo F, Di Gennaro E, Tatangelo F, Granata V, Cavalcanti E, Maiolino P, Bianco F, Aprea P, De Bellis M, Pecori B, Rosati G, Carlomagno C, Bertolini A, Gallo C, Romano C, Leone A, Caraco C, de Lutio di Castelguidone E, Daniele G, Catalano O, Botti G, Petrillo A, Romano GM, Iaffaioli VR, Lastoria S, Perrone F, Budillon A. A randomized phase 3 study on the optimization of the combination of bevacizumab with FOLFOX/OXXEL in the treatment of patients with metastatic colorectal cancer-OBELICS (Optimization of BEvacizumab scheduLIng within Chemotherapy Scheme). BMC Cancer. 2016 Feb 8;16:69. doi: 10.1186/s12885-016-2102-y. PMID 26857924

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Started | 115 | 115
Completed | 115 | 115
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [53 to 68] | 63 [56 to 68] | 62.3 [53.3 to 67.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 94
  Male | 69 | 67 | 136
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 115 | 115 | 230
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate (ORR), according to Response Evaluation Criteria in Solid Tumors (RECIST),version 1.1, was the primary end point and was defined as the number of complete plus partial responses divided by the number of enrolled patients.
  Per RECIST v 1.1 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Objective response was assessed by computed tomographic scan or other appropriate imaging at weeks 12 and 24 from randomization, and every 3 months thereafter, assessed up to 90 months.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Number analyzed (Participants) | 115 | 115
participants | 65 [47.0 to 65.7] | 66 [47.8 to 66.6]

2. Secondary Outcome: Disease Control Rate
Description: Disease control rate was calculated by adding complete and partial responses and stable disease.
Time Frame: At weeks 12 and 24 from randomization and every 3 months thereafter, assessed up to 90 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Number analyzed (Participants) | 115 | 115
Participants | 107 | 103

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to the date of death. Patients alive at the time of the final analysis were censored on the date of the last follow-up information available.
Time Frame: assessed up to 90 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Number analyzed (Participants) | 115 | 115
months | 29.8 [22.5 to 41.1] | 24.1 [18.6 to 29.8]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to the date of progression or death, whichever occurred first. Patients without progression were censored on the date of the last follow-up visit.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: assessed up to 90 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Number analyzed (Participants) | 115 | 115
months | 11.7 [9.9 to 12.9] | 10.5 [9.1 to 12.3]

5. Secondary Outcome: Toxic Effects
Description: Toxic effects were scored according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0. For the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE), version 4.0 scale score range from 1 to 4. A high score, that is 3 and 4, represents a high level of toxicity, whereas the minimum values, that is 1 and 2, represents a mild/modest level of toxicity.
Time Frame: up to 4 weeks after the end of the treatment
Population: any grade of toxic effects
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
Number analyzed (Participants) | 114 | 115
Participants | 108 | 113

ADVERSE EVENTS:
Time Frame: Evaluated every 2 weeks up to 6 months
Arm/Group | Bevacizumab Before Chemotherapy | Bevacizumab With Chemotherapy
All-Cause Mortality (participants affected / at risk) | 2/115 | 2/115
Serious Adverse Events (participants affected / at risk) | 65/115 | 75/115
Other Adverse Events (participants affected / at risk) | 108/115 | 113/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Before Chemotherapy (N=115) | Bevacizumab With Chemotherapy (N=115)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 19 (19)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Mucositis oral (Infections and infestations) | 4 (4) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (4) | 5 (5)
Fever (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2) | 4 (4)
Alanine aminotransferase level increased (Hepatobiliary disorders) | 1 (1) | 1 (1)
Alkaline phosphatase level increased (Hepatobiliary disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 23 (23) | 28 (28)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
White blood cell count decreased (Blood and lymphatic system disorders) | 5 (5) | 8 (8)
Peripheral neuropathy (Nervous system disorders) | 15 (15) | 15 (15)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Hypertension (Cardiac disorders) | 3 (3) | 7 (7)
Thromboembolic event (Vascular disorders) | 2 (2) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Before Chemotherapy (N=115) | Bevacizumab With Chemotherapy (N=115)
Anemia (Blood and lymphatic system disorders) | 28 (28) | 27 (27)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 27 (27) | 44 (44)
Mucositis oral (Infections and infestations) | 26 (26) | 34 (34)
Nausea (Gastrointestinal disorders) | 44 (44) | 44 (44)
Vomiting (Gastrointestinal disorders) | 6 (6) | 10 (10)
Fatigue (General disorders) | 16 (16) | 30 (30)
Fever (General disorders) | 8 (8) | 7 (7)
Pain (General disorders) | 5 (5) | 3 (3)
Allergic reaction (Immune system disorders) | 3 (3) | 4 (4)
Alanine aminotransferase level increased (Hepatobiliary disorders) | 23 (23) | 23 (23)
Alkaline phosphatase level increased (Hepatobiliary disorders) | 22 (22) | 23 (23)
Neutrophil count decreased (Blood and lymphatic system disorders) | 42 (42) | 44 (44)
Platelet count decreased (Blood and lymphatic system disorders) | 20 (20) | 32 (32)
White blood cell count decreased (Blood and lymphatic system disorders) | 28 (28) | 35 (35)
Peripheral neuropathy (Nervous system disorders) | 64 (64) | 70 (70)
Proteinuria (Renal and urinary disorders) | 10 (10) | 3 (3)
Epistaxis (Vascular disorders) | 15 (157) | 7 (7)
Voice alteration (General disorders) | 7 (7) | 6 (6)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (19) | 23 (23)
Hypertension (Cardiac disorders) | 32 (32) | 25 (25)
Thromboembolic event (Vascular disorders) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
Considering that the accuracy of conventional evaluation of tumor response by RECIST criteria to bevacizumab combination treatment has been questioned, we acknowledge that our choice of ORR as primary end point may have been inadequate.

We are also aware that balancing out unmeasurable differences in patient outcome through randomization is not always achieved with confidence in trials with a relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-10-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT01718873/Prot_SAP_000.pdf